CLINICAL TRIAL: NCT01696851
Title: Physiological and Psycho-social Variables of People With a Spinal Cord Injury
Brief Title: Physiological and Psycho-social Variables of People With a Spinal Cord Injury Participating in Competitive Rugby in Wheelchairs
Status: Withdrawn | Type: Observational
Why Stopped: no more interested in this issue
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-10-8276-GZ-CTIL
Record Dates: First submitted 2012-09-10; First posted 2012-10-01 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Wheelchair Rugby Players With Tetraplegia
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- wheelchair rugby players with tetraplegia
  Interventions: Other: tests and questionnaires
- other routine sport participants with tetraplegia
  Interventions: Other: tests and questionnaires

INTERVENTIONS:
Other: tests and questionnaires — lung test, depression and self-efficacy questionnaires and Functional testing.

SUMMARY:
People with Spinal cord injury with tetraplegia suffer from respiratory problem due to weakness of the muscles and because the autonomic system dysfunction.

Exercise is one way of preserving and improving physical fitness and directly and indirectly reduce risk factors such as insulin resistance, weight loss and low values of HDL. subjects with spinal cord injury with tetraplegia have limited options for exercise: table tennis, gym, pool and more. Because of the nature of the injury which includes the sympathetic failure, they can not easily get the desired pulse to improve physical fitness.

Wheelchair rugby in Canada was developed specifically for people with tetraplegia who could not participate in wheelchair basketball. The game combines short, quick races with different aerobic capabilities. Previous studies have shown that participants in wheelchair rugby Improve anaerobic power, oxygen consumption, physical fitness and daily functioning. Wheelchair rugby improves self-confidence and as a result it affects other areas of life. Another study examined sense of self-efficacy, saw improvement in this index for rugby players in a wheelchair at high levels.

In the present study the investigators aim to examine whether regular participation in wheelchair Rugby for a season has more impact than other routine exercise (table tennis, gym, swimming).

ELIGIBILITY:
Inclusion Criteria:

* subjects with tetraplegia who play wheelchair rugby

Exclusion Criteria:

* suffering from a medical condition that prevents from performing the tests required by the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Wheelchair rugby players with SCI with four limbs paralyzed playing and practicing regularly. Season lasts about six months.
  Belonging to this group are training and playing regularly twice a week about 3 hours at a time, total of 6 hours per week under the supervision of two coaches who attend every practice and game.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
lung function during rest using a spirometer | one minute
Functional testing | 5 minutes
  getting on a 6 meters long ramp adapted to the ability of people with tetraplegia (this takes up to 30 seconds). And opening and closing a sliding door.
Depression | 5 minutes
  Beck questionnaire assessing depression
Self efficacy | 5 minutes
  Sense of self efficacy questionnaire assessing self efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Gabi Zeilig, Dr., Principal Investigator — Sheba Medical Center
Locations (1):
- College of Physical Education Wingate, Netanya, Israel